CLINICAL TRIAL: NCT07207421
Title: The Effect of Ultra-Fast-Track Cardiac Anesthesia in Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Assoc. Prof., Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ADYU-ANS-NY-012
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft (CABG)
Keywords: Coronary Artery Bypass Graft (CABG); ultra- fast track anesthesia; Vaso-Inotropic Score (VIS); Postoperative recovery; Cardiac anesthesia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, controlled, parallel assignment trial with two groups. Participants undergoing elective coronary artery bypass grafting (CABG) will be randomized in a 1:1 ratio to either Ultra-Fast-Track anesthesia with early extubation (intervention group) or standard extubation in the intensive care unit (control group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-Fast-Track Anesthesia group (Experimental): Patients will receive standard general anesthesia for cardiac surgery. Extubation will be targeted in the operating room or within the first postoperative hour before ICU transfer.
  Interventions: Procedure: Ultra-Fast-Track Anesthesia
- Standard care group (Active Comparator): Patients will receive standard general anesthesia for cardiac surgery. They will remain intubated upon ICU admission and will be extubated according to routine ICU protocols.
  Interventions: Procedure: Standart care anesthesia

INTERVENTIONS:
Procedure: Ultra-Fast-Track Anesthesia — General anesthesia for cardiac surgery followed by planned extubation in the operating room or within the first postoperative hour before ICU transfer.
  Arms: Ultra-Fast-Track Anesthesia group
Procedure: Standart care anesthesia — Extubation will be targeted in the ICU according to respiratory effort.
  Arms: Standard care group

SUMMARY:
This randomized controlled trial aims to evaluate the impact of Ultra-Fast-Track (UFT) anesthesia on postoperative recovery in patients undergoing elective coronary artery bypass grafting (CABG). UFT anesthesia targets extubation in the operating room or within the first hour after surgery, whereas standard care involves transfer to the intensive care unit (ICU) with subsequent extubation according to routine protocols. A total of 100 patients will be randomized in a 1:1 ratio. The primary outcome is the maximum Vaso-Inotropic Score (VIS) within the first 24 postoperative hours. Secondary outcomes include postoperative pain scores (VAS), Quality of Recovery-15 (QoR-15) scores, opioid and analgesic requirements, ICU and hospital length of stay, time to mobilization, and postoperative complications. This study seeks to determine whether UFT anesthesia can safely reduce inotropic support requirements and enhance early recovery following CABG.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is the most frequently performed cardiac surgical procedure and remains the gold standard for the treatment of advanced coronary artery disease. While CABG restores myocardial perfusion and relieves ischemic symptoms, the postoperative period is often associated with prolonged mechanical ventilation, increased risk of complications, higher costs, and delayed recovery.

Ultra-Fast-Track (UFT) anesthesia is a perioperative strategy that aims to achieve extubation either in the operating room or within the first postoperative hour. Previous studies have demonstrated that fast-track and UFT protocols may shorten intensive care unit (ICU) length of stay, reduce postoperative complications, and improve recovery, without compromising patient safety. However, the influence of UFT anesthesia on inotropic support requirements, recovery quality, and analgesic needs in patients undergoing CABG has not been fully clarified.

In this prospective, randomized, controlled clinical trial, 100 patients scheduled for elective CABG will be randomly assigned to one of two groups:

UFT group: patients will undergo standard general anesthesia for cardiac surgery and will be extubated in the operating room or within one hour postoperatively before ICU transfer.

Standard care group: patients will undergo the same anesthesia protocol but will remain intubated upon ICU admission, with extubation performed according to routine ICU protocols.

The primary endpoint is the maximum Vaso-Inotropic Score (VIS) recorded during the first 24 hours after surgery. Secondary endpoints include postoperative pain scores (VAS), opioid and analgesic requirements, Quality of Recovery-15 (QoR-15) scores at 24 and 72 hours, ICU and hospital length of stay, time to mobilization, and the incidence of postoperative complications such as reintubation, pneumonia, atrial fibrillation, and acute kidney injury.

This study is designed to provide high-quality evidence on whether UFT anesthesia can safely decrease inotropic support requirements, enhance postoperative recovery, and reduce ICU stay in patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years undergoing elective coronary artery bypass grafting (CABG)
* Patients suitable for Ultra-Fast-Track anesthesia as determined by the anesthesia team
* Ability to provide written informed consent

Exclusion Criteria:

* Emergency CABG or combined cardiac procedures (e.g., valve surgery)
* Preoperative shock or requirement for mechanical ventilation
* Severe pulmonary disease (e.g., GOLD stage 3-4 COPD, home oxygen therapy)
* Severe hepatic failure or end-stage renal disease requiring dialysis
* Pregnancy
* Inability to provide informed consent or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Vaso-Inotropic Score (VIS) | From the end of surgery (0 hour) up to 24 hours postoperatively, with hourly assessments
  The Vaso-Inotropic Score (VIS) will be calculated hourly based on recorded inotrope and vasopressor infusion rates using the standard VIS calculation method. The primary outcome is the maximum (peak) VIS value observed during the first 24 postoperative hours. VIS values will be extracted from infusion charts and/or electronic medical records.

SECONDARY OUTCOMES:
Quality of Recovery (QoR-15) score | 24 hour postoperatively
  Assessed using the validated QoR-15 questionnaire to evaluate patient-reported recovery, including physical comfort, emotional state, and pain.
Postoperative pain score (VAS) | Postoperative 2, 4, 6, 8, 12, and 24 hours (within the first 24 hours after surgery)
  Visual Analog Scale (VAS); range: 0-10, where higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Training and Research Hospital, Adıyaman, Adıyaman Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided